CLINICAL TRIAL: NCT03995108
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of Mavorixafor in Patients With WHIM Syndrome With Open-Label Extension
Brief Title: Efficacy and Safety Study of Mavorixafor in Participants With Warts, Hypogammaglobulinemia, Infections, and Myelokathexis (WHIM) Syndrome
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: X4 Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: X4P-001-103; 2019-001153-10 (EudraCT Number); 4WHIM (Other: X4 Pharmaceuticals)
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: WHIM Syndrome
MeSH Terms: conditions — WHIM syndrome | interventions — mavorixafor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mavorixafor (Experimental): Participants (adults and adolescents [12 to 17 years of age weighing >50 kilograms [kg]) will receive mavorixafor 400 milligrams (mg) once daily (QD) orally for 52 weeks in the Randomized Placebo-Controlled Period. Adolescents weighing ≤50 kg will receive mavorixafor 200 mg QD. Participants who complete the Randomized Placebo-Controlled Period or are granted Early Release due to recurrent or significant infections, as adjudicated by a blinded, independent adjudication committee (AC), will be offered the opportunity to enroll in the Open-Label Period and receive treatment with mavorixafor 400 mg once daily orally until commercial availability or study termination by the Sponsor.
  Interventions: Drug: Mavorixafor
- Placebo (Placebo Comparator): Participants will receive placebo matching to mavorixafor QD orally for 52 weeks in the Randomized Placebo-Controlled Period. Participants who complete the Randomized Placebo-Controlled Period or are granted Early Release due to recurrent or significant infections, as adjudicated by a blinded, independent AC, will be offered the opportunity to enroll in the Open-Label Period and receive treatment with mavorixafor 400 mg once daily orally until commercial availability or study termination by the Sponsor.
  Interventions: Drug: Mavorixafor; Drug: Placebo

INTERVENTIONS:
Drug: Mavorixafor — Mavorixafor provided as 100 mg capsules.
  Other Names: AMD11070; X4P-001
Drug: Placebo — Placebo matching to mavorixafor capsules
  Arms: Placebo

SUMMARY:
This study has a double-blind, Randomized Placebo-Controlled Period and an Open-Label Period. The primary objective of the Randomized Placebo-Controlled Period is to demonstrate the efficacy of mavorixafor in participants with WHIM syndrome as assessed by increasing levels of circulating neutrophils compared with placebo, and relative to a clinically meaningful threshold. The primary objective of the Open-Label Period is to evaluate the safety and tolerability of mavorixafor in participants with WHIM syndrome. Participants are allowed to continue treatment in the Open-Label Period, if regionally applicable, until mavorixafor becomes commercially available, or until the study is terminated by the Sponsor.

ELIGIBILITY:
Inclusion Criteria for the Randomized Placebo-Controlled Period :

* Have signed the current approved informed consent form. Participants under 18 years of age (in the Netherlands and other applicable regions, participants under 16 years of age) will sign an approved informed assent form and must also have a signed parental/legal guardian consent.
* Have a genotype-confirmed mutation of chemokine (C-X-C motif) receptor 4 (CXCR4) consistent with WHIM phenotype.
* Agree to use a highly effective form of contraception.
* Be willing and able to comply with the protocol.
* Have confirmed ANC ≤400 cells/µL during screening, obtained while participant has no clinical evidence of infection.

Inclusion Criteria for the Open-Label Period:

* Completed the Randomized Period; or
* Granted Early Release from the Randomized Period.

Exclusion Criteria:

* Has known systemic hypersensitivity to the mavorixafor drug substance, its inactive ingredients, or the placebo.
* Is pregnant or breastfeeding.
* Has any medical or personal condition, which in the opinion of the Investigator may potentially compromise the safety or compliance of the participant or may preclude the participant's successful completion of the clinical study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Randomized Placebo-Controlled Period: Time (in Hours) Above Threshold-Absolute Neutrophil Count (TAT-ANC in hours) of ≥ 500 Cells/Microliter (µL) over a 24-hour period | Time 0 (pre-dose, up to 15 minutes prior), 30, 60, and 90 min (each ± 5 min) and 2, 3, 4, 8, 12, 16, and 24 hours (each ± 15 min) post-dose at Baseline, Weeks 13, 26, 39, and 52
Open-Label Period: Percentage of Participants With Adverse Events (AEs) | From Day 1 (end of randomized period) up to end of study (30 days post-treatment in open-label period [Week 56 of open-label period])

SECONDARY OUTCOMES:
Randomized Placebo-Controlled Period: Time (in Hours) Above Threshold-Absolute Lymphocyte Count (TAT-ALC) of ≥ 1000 Cells/µL over a 24-hour period | Time 0 (pre-dose, up to 15 minutes prior), 30, 60, and 90 minutes (each ± 5 minutes) and 2, 3, 4, 8, 12, 16, and 24 hours (each ± 15 minutes) post-dose at Baseline, Weeks 13, 26, 39, and 52
Randomized Placebo-Controlled Period: Composite Clinical Efficacy for Mavorixafor based on total infection score and total wart change score | Baseline up to Week 52
Randomized Placebo-Controlled Period: Change From Baseline in Total Warts Score at Week 52 | Baseline, Week 52
Randomized Placebo-Controlled Period: Total Infection Score for Mavorixafor | Baseline up to Week 52
Randomized Placebo-Controlled Period: Time to Early Release | Baseline up to Week 52
Randomized Placebo-Controlled Period: TAT-ALC of ≥ 1000 Cells/µL in Participants With Lymphopenia | Baseline
Randomized Placebo-Controlled Period: Total Infection Score for Participants With Non-Immunoglobulin (non-Ig) Use (Percentage of Participants With Infections) | Baseline up to Week 52
Randomized Placebo-Controlled Period: Change in Total Wart Score at Baseline, Based on Clinical Global Impression of Change (CGI-C) | Baseline
Randomized Placebo-Controlled Period: Composite Clinical Efficacy (Total Infection Score and Total Wart Change Score) for Participants With Non-Ig Use | Baseline up to Week 52
  Composite clinical efficacy will be calculated using the total infection score and total wart change score for participants with warts at baseline or non-Ig use. It will be analyzed by a blinded, independent AC.
Randomized Placebo-Controlled Period: Change in Total Wart Score at Baseline (CGI-C), Based on Local Dermatologist Review | Baseline
Randomized Placebo-Controlled Period: Participant Global Impression of Change (PGI-C) | Baseline up to Week 52
Randomized Placebo-Controlled Period: Participant Global Impression of Severity (PGI-S) | Baseline up to Week 52
Randomized Placebo-Controlled Period: Vaccine Titer Levels at Week 52 in Participants Vaccinated at Week 13, With Tetanus, Diphtheria, and Pertussis (Tdap) Including Pertussis Toxin, and Tetanus | Week 52
Randomized Placebo-Controlled Period: Vaccine Titer Levels at Week 52 for Human Papillomavirus (HPV) 16 and HPV 18 in Participants Receiving Vaccinations With HPV 9-Valent Vaccine, Recombinant (Gardasil®9) | Week 52
Randomized Placebo-Controlled Period: Change From Baseline in Clinical Global Impression of Severity (CGI-S), Based on Local Dermatologist Review | Baseline up to Week 52
Randomized Placebo-Controlled Period: Number of Participants with Infections | Baseline up to Week 52
Randomized Placebo-Controlled Period: Infection-Free Time | Baseline up to Week 52
Randomized Placebo-Controlled Period: Number of Days Lost From Work/School | Baseline up to Week 52
Randomized Placebo-Controlled Period: Quality of Life as Measured by 36-Item Short Form Survey Score | Baseline up to Week 52
Randomized Placebo-Controlled Period: Quality of Life as Measured by EuroQoL-5 Dimension-5 Level (EQ-5D-5L) Score | Baseline up to Week 52
Randomized Placebo-Controlled Period: Quality of Life as Measured by Life Quality Index (LQI) Score | Baseline up to Week 52
Randomized Placebo-Controlled Period: Quality of Life as Measured by Dermatology LQI Score | Baseline up to Week 52
Randomized Placebo-Controlled Period: Quality of Life as Measured by Pediatric Quality of Life Inventory (PedsQL) Score | Baseline up to Week 52
Randomized Placebo-Controlled Period: Change From Baseline in Anogenital (AG) Warts Based on Dermatologist CGI-C Assessment | Baseline to Week 52
Randomized Placebo-Controlled Period: Change From Baseline in Anogenital (AG) Warts Based on AG Wart Severity Assessment | Baseline to Week 52
Randomized Placebo-Controlled Period: Number of Events Requiring Rescue Treatment Due to Infection | Baseline to Week 52
Randomized Placebo-Controlled Period: Number of Participants With Incidence and Duration of Hospitalizations Due to Infection | Baseline to Week 52
Randomized Placebo-Controlled Period: Number of Participants With Incidence of Newly Developed Warts | Baseline to Week 52
Randomized Placebo-Controlled Period: Area Under the Curve for ANC (AUCANC) Using Trapezoidal Method | Time 0 (pre-dose, up to 15 minutes prior), 30, 60, and 90 minutes (each ± 5 minutes) and 2, 3, 4, 8, 12, 16, and 24 hours (each ± 15 minutes) post-dose at Baseline, Weeks 13, 26, 39, and 52
Randomized Placebo-Controlled Period: Percentage of Neutrophil Responders | Baseline up to Week 52
Randomized Placebo-Controlled Period: Mavorixafor Treatment Group: AUCANC | Time 0 (pre-dose, up to 15 minutes prior), 30, 60, and 90 minutes (each ± 5 minutes) and 2, 3, 4, 8, 12, 16, and 24 hours (each ± 15 minutes) post-dose at Baseline, Weeks 13, 26, 39, and 52
Randomized Placebo-Controlled Period: Area Under the Curve for ALC (AUCALC) | Time 0 (pre-dose, up to 15 minutes prior), 30, 60, and 90 minutes (each ± 5 minutes) and 2, 3, 4, 8, 12, 16, and 24 hours (each ± 15 minutes) post-dose at Baseline, Weeks 13, 26, 39, and 52
Randomized Placebo-Controlled Period: Percentage of Lymphocyte Responders | Baseline up to Week 52
Randomized Placebo-Controlled Period: Change From Baseline in Total ALC, Absolute Monocyte Count (AMC), ANC, and White Blood Cell (WBC) at Week 52 | Baseline, Week 52
Absolute and Fold Change From Baseline in Absolute T, B and Natural Killer Lymphocyte at Week 52 | Baseline, Week 52
Randomized Placebo-Controlled Period: Number of Participants With AEs | Baseline up to Week 52
Randomized Placebo-Controlled Period: Pharmacokinetics (PK), Maximum Observed Plasma Concentration (Cmax) of Mavorixafor | Time 0 (pre-dose, up to 15 minutes prior), 30, 60, and 90 minutes (each ± 5 minutes) and 2, 3, 4, 8, 12, 16, and 24 hours (each ± 15 minutes) post-dose at Weeks 13, 26, 39, and 52; and 4 hours post-dose at Baseline
Randomized Placebo-Controlled Period: PK, Time to Reach Cmax (Tmax) of Mavorixafor | Time 0 (pre-dose, up to 15 minutes prior), 30, 60, and 90 min (each ± 5 minutes) and 2, 3, 4, 8, 12, 16, and 24 hours (each ± 15 minutes) post-dose at Weeks 13, 26, 39, and 52; and 4 hours post-dose at Baseline
Randomized Placebo-Controlled Period: PK, Half-Life of (T1/2) of Mavorixafor | Time 0 (pre-dose, up to 15 minutes prior), 30, 60, and 90 minutes (each ± 5 minutes) and 2, 3, 4, 8, 12, 16, and 24 hours (each ± 15 minutes) post-dose at Weeks 13, 26, 39, and 52; and 4 hours post-dose at Baseline
Randomized Placebo-Controlled Period: PK, Area Under the Curve (AUC) of Mavorixafor | Time 0 (pre-dose, up to 15 minutes prior), 30, 60, and 90 minutes (each ± 5 minutes) and 2, 3, 4, 8, 12, 16, and 24 hours (each ± 15 minutes) post-dose at Weeks 13, 26, 39, and 52; and 4 hours post-dose at Baseline
Open-Label Period: Percentage of Neutrophil Responders | Baseline up to Week 52 of open-label period
Open-Label Period: Percentage of Lymphocyte Responders | Baseline up to Week 52 of open-label period
Open-Label Period: Absolute and Fold Change From Baseline in Total ALC, AMC, ANC, and WBC at Week 52 | Baseline up to Week 52 of open-label period
Open-Label Period: Vaccine Titer Levels During the First Year of Open-Label Period, in Participants Vaccinated With Tdap During the Study Including Pertusis Toxin and Tetanus | Year 1 of open-label period
Open-Label Period: Vaccine Titer Levels During the First Year of the Open-Label Period for HPV 16 and HPV 18 in Participants Receiving Vaccinations With HPV 9-Valent Vaccine, Recombinant (Gardasil®9) During the Study | Year 1 of open-label period
Open-Label Period: Change From Baseline in Cutaneous Warts at Week 52, Based on Central Review of CGI-C | Baseline, Week 52 of open-label period
Open-Label Period: Change From Baseline in Cutaneous Warts, Based on Central Review of CGI-S | Baseline, Week 52 of open-label period
Open-Label Period: Change From Baseline in Cutaneous Warts, Based on Local Dermatologist CGI-C | Baseline, Week 52 of open-label period
Open-Label Period: Change From Baseline in Cutaneous Warts, Based on Local Dermatologist CGI-S | Baseline, Week 52 of open-label period
Open-Label Period: Change Over Time in PGI-C | Baseline up to Week 52 of open-label period
Open-Label Period: Change Over Time in PGI-S | Baseline up to Week 52 of open-label period
Open-Label Period: Total Infection Score (Percentage of Participants With Infections) | Baseline up to Week 52 of open-label period

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — X4 Pharmaceuticals
Locations (23):
- United States (6):
  - University of California San Diego Health/Rady Children's Hospital, San Diego, California
  - California Dermatology Institute, Thousand Oaks, California
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University Medical Center, Baltimore, Maryland
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Washington Medical Center, Seattle, Washington
- Australia (2):
  - Wesley Hospital, Auchenflower, Queensland
  - Children's Health Queensland Hospital, South Brisbane, Queensland
- Medical University of Vienna - Medizinische Universität Wien, Vienna, Austria
- Aarhus University Hospital, Aarhus, Denmark
- France (3):
  - CHU de Lyon, Institut d'Hematologie et d'Oncologie Pediatrique, Lyon, Rhne
  - CHU Paris Est, Hôpital d'Enfants Armand-Trousseau, Paris
  - Hopital Necker-Enfants Malades, Paris
- University of Debrecen, Affiliated Department of Infectology, Debrecen, Hajdú-Bihar, Hungary
- HaEmek Medical Center, Afula, Israel
- Università degli Studi di Brescia, Scienze Cliniche e Sperimentali, Brescia, Piazza Del Mercato, Italy
- Emma Children's Hospital Academic Medical Center (AMC), Amsterdam, Netherlands
- Russia (2):
  - Dmitry Rogachev National Research Center of Pediatric Hematology, Oncology and Immunology, Moscow
  - Academician I.P. Pavlov First Saint Petersburg State Medical University, Saint Pertersburg
- Seoul National University Hospital, Children's Hospital, Seoul, South Korea
- Spain (2):
  - Hospital Sant Joan de Deu Barcelona, Barcelona, Esplugues de Llobregat
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
- Cukurova University Faculty of Medicine, Sarıçam, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Badolato R, Alsina L, Azar A, Bertrand Y, Bolyard AA, Dale D, Deya-Martinez A, Dickerson KE, Ezra N, Hasle H, Kang HJ, Kiani-Alikhan S, Kuijpers TW, Kulagin A, Langguth D, Levin C, Neth O, Olbrich P, Peake J, Rodina Y, Rutten CE, Shcherbina A, Tarrant TK, Vossen MG, Wysocki CA, Belschner A, Bridger GJ, Chen K, Dubuc S, Hu Y, Jiang H, Li S, MacLeod R, Stewart M, Taveras AG, Yan T, Donadieu J. A phase 3 randomized trial of mavorixafor, a CXCR4 antagonist, for WHIM syndrome. Blood. 2024 Jul 4;144(1):35-45. doi: 10.1182/blood.2023022658. PMID 38643510